CLINICAL TRIAL: NCT07129278
Title: Breathwork Intervention for Individuals With Post-Traumatic Stress Symptoms
Brief Title: Breathwork Intervention for Posttraumatic Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Licensed Psychologist and an Associate Professor, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005111
Record Dates: First submitted 2025-04-30; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: PTSD
Keywords: PTSD; Breathwork; Contemplative practice; Cyclic sighing
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Treatment (Experimental): All participants will be assigned to breathwork.
  Interventions: Behavioral: Breathwork

INTERVENTIONS:
Behavioral: Breathwork — Participants will complete their single-session, 2-hour training in a small group with the Breathwork instructor.

SUMMARY:
The goal of this single-site, single-arm pilot study is to examine the impact of breathwork training for posttraumatic stress symptoms in an adult veteran population. Participants will complete a single, in-person breathwork session (2 hours) led by a certified breathwork facilitator and engage in an integration session (30 minute) with a licensed psychologist. Participants will be invited to engage in two, optional, virtual follow up breathwork sessions (40 minute practice each) during weeks 2 and 3 following the in-person breathwork session.

ELIGIBILITY:
Inclusion Criteria:

* (1) having received a professional diagnosis of post-traumatic stress disorder (PTSD)
* (2) being able not to commit to another (new) treatment during the course of the study
* (3) understanding English instructions fluently
* (4) being 18 and above.

Exclusion Criteria:

* (1) having been exposed to breathwork any time in the past
* (2) being unable to perform most basic tasks due to PTSD or other mental illness.
* (3) Asthma, breathing problems, or a respiratory disorder (e.g., chronic obstructive pulmonary disease).
* (4) Uncontrolled hypertension (i.e., systolic blood pressure/diastolic blood pressure > 150/95), orthostatic hypotension (e.g., issues with fainting), or cardiovascular or peripheral arterial disease.
* (5) Current or past diagnosis of a neurological disease (e.g., Parkinson's, multiple sclerosis, epilepsy, vasovagal syncope)
* (6) Serious psychiatric disorder requiring hospitalization within the past 12 months
* (7) Current substance use disorder or history of hospitalization for treatment of a substance use disorder.
* (8) Current participation in another research study involving an intervention or treatment.
* (9) Currently pregnant
* (10) Any significant comorbidities or issues that, in the opinion of the investigators, could interfere with the study or lead to deleterious effects for the participant.
* (11) Adults unable to consent
* (12) Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | From date of first participant contact (May 6th) to the day before the final breathwork session (10th of October): 158 days
  The primary outcome of recruitment feasibility will be assessed by the ability to enroll 30 eligible participants by September 30, 2025. This will inform the practicality of recruitment strategies for a future definitive trial.
Retention | From baseline assessment (-2 weeks) to 13-week follow-up: 15 week span
  ≥80% of enrolled participants completing all study procedures through final follow-up.
Acceptability of Intervention Measure (AIM) | Administered once at the conclusion of the in-person integration session (approx. 30 minutes post-intervention)
  Acceptability of Intervention Measure (AIM) is a 4-item scale. It uses a 5-point ordinal scale for each item, ranging from "Completely Disagree" to "Completely Agree". Scores are typically calculated as either the mean or total of the responses, with higher scores indicating greater acceptability.
Intervention Appropriateness Measure (IAM) | Administered once at the conclusion of the in-person integration session (approx. 30 minutes post-intervention)
  Intervention Appropriateness Measure (IAM) is a 4-item scale. It uses a 5-point ordinal scale for each item, ranging from "Completely Disagree" to "Completely Agree". Scores are typically calculated as either the mean or total of the responses, with higher scores indicating greater appropriateness.
Feasibility of Intervention Measure (FIM) | Administered once at the conclusion of the in-person integration session (approx. 30 minutes post-intervention)
  Feasibility of Intervention Measure (FIM) is a 4-item scale. It uses a 5-point ordinal scale for each item, ranging from "Completely Disagree" to "Completely Agree". Scores are typically calculated as either the mean or total of the responses, with higher scores indicating greater feasibility.
Acupuncture Expectancy Scale (AES) | Administered once at the conclusion of the in-person integration session (approx. 30 minutes post-intervention)
  The Acupuncture Expectancy Scale (AES) is a 4-item scale. It uses a 5-point Likert scale for each item, and a higher total score (ranging from 4 to 20) indicates greater expectancy of benefit from acupuncture.

SECONDARY OUTCOMES:
Post-Traumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Baseline (-2 weeks), 4-week follow up, 8-week follow up and 13-week follow-up: 15 week span
  The PCL-5 is a 20-item self-report measure. It is scored by summing the ratings for each of the 20 items. Each item is rated on a 5-point scale (0-4), where 0 means "Not at all" and 4 means "Extremely". The total score, ranging from 0 to 80, represents the severity of PTSD symptoms.
Brief Trauma Questionnaire (BTQ) | Baseline (-2 weeks), 4-week follow up, 8-week follow up and 13-week follow-up: 15 week span
  The BTQ is a 10-item instrument that lists a number of difficult of stressful things that sometimes happen to people. The Brief Trauma Questionnaire (BTQ) is scored by counting the number of traumatic events experienced that meet DSM-IV "Criterion A" criteria (life threat or serious injury). Each of the 10 items on the BTQ is scored as positive if the respondent reports experiencing the event and also reports either life threat or serious injury (depending on the specific question). A higher score indicates a greater number of traumatic events experienced
Posttraumatic Growth Inventory (PGI) | Baseline (-2 weeks), 4-week follow up, 8-week follow up and 13-week follow-up: 15 week span
  Posttraumatic growth will be assessed with the 21-item Posttraumatic Growth Inventory (PGI). It is scored by summing responses to its 21 items, each rated on a 6-point Likert scale. The total score ranges from 0 to 105, with higher scores indicating greater perceived post-traumatic growth. Scores on the five subscales (Relating to Others, New Possibilities, Personal Strength, Spiritual Change, and Appreciation of Life) are calculated by averaging the relevant items within each subscale.
Patient Health Questionnaire 2-item (PHQ-2) | Baseline; 2-week follow up; 6-week follow up.
  The Patient Health Questionnaire 2-item (PHQ-2) is scored by summing the responses to its two questions. Each question offers four possible responses, scored from 0 to 3, with 0 being "not at all" and 3 being "nearly every day". A total score is calculated by adding the scores of both questions, resulting in a range from 0 to 6. A score of 3 or higher suggests further evaluation for depression
Generalized Anxiety Disorder-2 (GAD-2) | Baseline (-2 weeks), 4-week follow up, 8-week follow up and 13-week follow-up: 15 week span
  Patients will note their anxiety with the Generalized Anxiety Disorder-2 (GAD-2). This 2-item scale is scored by summing the responses to two questions, each rated on a 4-point scale. The possible scores for each item range from 0 to 3, with 0 representing "Not at all" and 3 representing "Nearly every day". The total score, which ranges from 0 to 6, is then calculated by adding the scores of the two items. A higher score indicates a greater likelihood of anxiety.
Pain, Enjoyment of Life, and General Activity Scale (PEG) | Baseline (-2 weeks), 4-week follow up, 8-week follow up and 13-week follow-up: 15 week span
  Participants will be asked about their pain intensity and pain interference with the Pain, Enjoyment of Life and General Activity (PEG) Scale. The 11-item Likert scale is scored by averaging the responses to three questions, each rated on a scale of 0 to 10. A higher score indicates a greater impact of pain.
PROMIS Sleep Disturbance 6a + Sleep Duration | Baseline (-2 weeks), 4-week follow up, 8-week follow up and 13-week follow-up: 15 week span
  The PROMIS Sleep Disturbance 6a and Sleep Duration measures are scored by first summing the responses to the individual items, then converting the raw sum score to a standardized T-score using conversion tables. The PROMIS Sleep Disturbance 6a uses a 5-point Likert scale for each item, and the Sleep Duration is a separate item with its own scoring. The T-score represents the individual's sleep disturbance relative to a reference population (mean of 50, standard deviation of 10).
PROMIS v1.0 Alcohol Use - Short Form 7a | Baseline (-2 weeks), 4-week follow up, 8-week follow up and 13-week follow-up: 15 week span
  The PROMIS v1.0 Alcohol Use - Short Form 7a is a 7-item questionnaire using a 5-point Likert scale (1- never to 5- almost always). It is scored by summing the responses to each question, where each question has a 5-point Likert scale. Higher scores indicate stronger positive expectancies about alcohol use. The raw score is then converted to a T-score for comparison with a normative sample.
Smoking: Nicotine Dependence for All Smokers - Short Form 4a | Baseline (-2 weeks), 4-week follow up, 8-week follow up and 13-week follow-up: 15 week span
  The Smoking: Nicotine Dependence for All Smokers - Short Form 4a is a 4-item questionnaire using a 5-point Likert scale (1-never, 5-always). The Smoking: Nicotine Dependence for All Smokers - Short Form 4a is scored by summing the values of the responses to each of its four items. Each item has five possible response options, ranging from 1 to 5, with higher scores indicating greater nicotine dependence. The total raw score ranges from 4 (lowest dependence) to 20 (highest dependence).
Patient Global Impression of Change (PGIC) | Baseline (-2 weeks), 4-week follow up, 8-week follow up and 13-week follow-up: 15 week span
  The PGIC is a single-item, seven-point scale used to assess a patient's perception of change in their condition since a specific point in time. The scale ranges from "very much worse" to "very much improved". Higher scores indicate greater improvement, while lower scores indicate worsening or no change.
Nondual Awareness Dimensional Assessment (NADA-State) | From immediately before to immediately after the in-person breathwork session (approximately 2-hour span); and from immediately before to immediately after each optional virtual follow-up session.
  Participants will complete the 3-item, state version of the Nondual Awareness Dimensional Assessment. The NADA is scored 0-10 and responses are averaged across the 3-items. A higher score is indicative of a greater self-transcendent state.
Emotional Breakthrough Inventory (EBI) | From immediately before to immediately after the in-person breathwork session (approximately 2-hour span); and from immediately before to immediately after each optional virtual follow-up session.
  The Emotional Breakthrough Inventory is a 6-item questionnaire to assess emotional breakthrough resulting from an experience. It is scored 0-10 and scores are summed, with a higher score being indicative of a greater emotional breakthrough.
Perceived Body Boundary Scale (PBBS) | From immediately before to immediately after the in-person breathwork session (approximately 2-hour span); and from immediately before to immediately after each optional virtual follow-up session.
  The Perceived Body Boundary Scale is a single visual item used to assess the strength of the boundary between the self and the world using a 7-point Likert type scale (1=Weak boundary, 7=Strong boundary).
Spatial Frame of Reference Continuum (SFoRC) | From immediately before to immediately after the in-person breathwork session (approximately 2-hour span); and from immediately before to immediately after each optional virtual follow-up session.
  The single-item Spatial Frame of Reference Continuum describes a spectrum of ways individuals and organisms represent and interact with spatial information, ranging from response A (self-centered (egocentric)) to response G (world-centered (allocentric) perspectives). Response G indicates the highest level of world-centered perspective.
Inclusion of Other in Self Scale (IOS) | From immediately before to immediately after the in-person breathwork session (approximately 2-hour span); and from immediately before to immediately after each optional virtual follow-up session.
  The Inclusion of Other in Self (IOS) is a single-item scale. It is scored by having the respondent select one of seven pairs of overlapping circles that best represents their relationship with another person or group. Each pair of circles represents a different level of overlap, from completely separate (1) to almost completely overlapping (7). The chosen number (1-7) serves as the score, indicating the degree of perceived closeness and interconnectedness.
Nondual Awareness Dimensional Assessment-Trait (NADA-T) | From immediately before to immediately after the in-person breathwork session (approximately 2-hour span); and from immediately before to immediately after each optional virtual follow-up session.
  The 13-item Nondual Awareness Dimensional Assessment-Trait (NADA-T) will be used to assess traits of consciousness. The Nondual Awareness Dimensional Assessment-Trait (NADA-T) is scored by summing responses to 13 items, each on a 5-point Likert scale, ranging from "never or very rarely" to "very often or always". The scale assesses two dimensions of nondual awareness: self-transcendence and bliss. The total score can range from 13 to 65, with higher scores indicating a greater experience of nondual awareness.
Integration Engagement Scale (IES) | 4-week follow up, 8-week follow up and 13-week follow-up
  The Integration Engagement Scale is a 12-item questionnaire used to measure positive behavioral engagement with integration. Participants are asked to rate their experiences on a 5-point Likert scale (0 = not at all to 4 = extremely). The IES yields a total score, typically ranging from 0 to 60. Higher scores on the IES generally indicate increased positive behavioral engagement with integration.
Experienced Integration Scale (EIS) | 4-week follow up, 8-week follow up and 13-week follow-up
  The Experienced Integration Scale is a 12-item questionnaire to capture internal aspects of feeling integrated. Participants are asked to rate their experiences on a 5-point Likert scale (1- strongly disagree to 5=strongly agree). Items are summed; a higher score indicates greater feelings of integration.
Whole Person Health Index | 4-week follow up, 8-week follow up and 13-week follow-up
  The Whole Person Health Index (WPHI) is a 9-item survey. It is scored by The WPHI can be calculated by summing the nine response scores, such that, over time, for example, an individual's WPHI going from 45 to 25 would indicate an improvement in overall self-assessed health
Brief Inventory of Psychosocial Functioning (B-IPF) | Baseline (-2 weeks), 4-week follow up, 8-week follow up and 13-week follow-up: 15 week span
  Psychosocial functioning will be assessed using the Brief Inventory of Psychosocial Functioning (B-IPF), a validated 7-item self-report instrument designed to measure psychosocial impairment across key life domains. Each item is rated on a 7-point Likert scale ranging from 0 ("Not at all") to 6 ("Very much"), with higher scores indicating greater psychosocial impairment. The total score is calculated by summing responses across all items, yielding a possible range of 0 to 42.
  Sample item: "I had trouble in my romantic relationship with my spouse or partner.
Single-Item State Anxiety Measure | From immediately before to immediately after the in-person breathwork session (approximately 2-hour span); and from immediately before to immediately after each optional virtual follow-up session.
  State anxiety will be measured using a single item adapted from the Generalized Anxiety Disorder 2-item (GAD-2) scale: "Right now, to what extent are you feeling… nervous, anxious, or on edge?" Participants respond using a 7-point Likert scale ranging from 0 ("Not at all") to 6 ("Extremely"), with higher scores indicating greater state anxiety.
Single-Item State Optimism Measure | From immediately before to immediately after the in-person breathwork session (approximately 2-hour span); and from immediately before to immediately after each optional virtual follow-up session.
  State optimism will be assessed using a single item adapted from the State Optimism Measure: "Right now, to what extent are you feeling… optimistic about life's challenges?" Participants respond using a 7-point Likert scale ranging from 0 ("Not at all") to 6 ("Extremely"), with higher scores indicating greater state optimism.
Single-Item State Relaxation Measure | From immediately before to immediately after the in-person breathwork session (approximately 2-hour span); and from immediately before to immediately after each optional virtual follow-up session.
  State relaxation will be measured using a single item adapted from the Relaxation State Questionnaire: "Right now, to what extent are you feeling… refreshed and awake?" Participants respond using a 7-point Likert scale ranging from 0 ("Not at all") to 6 ("Extremely"), with higher scores indicating greater relaxation or alertness.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Diamond Rose Sanctuary, Branford, Connecticut
  - Florida State University, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with qualified researchers upon request.

DOCUMENTS (1):
  • Informed Consent Form (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT07129278/ICF_000.pdf